CLINICAL TRIAL: NCT01082211
Title: A Phase II Study of Repeat Breast Preserving Surgery and 3D-Conformal Partial Breast Re-Irradiation (PBrI) for Local Recurrence of Breast Carcinoma
Brief Title: Radiation Therapy in Treating Women With Locally Recurrent Breast Cancer Previously Treated With Repeat Breast-Preserving Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RTOG 1014; CDR0000666991
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Breast Cancer
Keywords: invasive ductal breast carcinoma; medullary ductal breast carcinoma with lymphocytic infiltrate; invasive lobular breast carcinoma; tubular ductal breast carcinoma; mucinous ductal breast carcinoma; ductal breast carcinoma in situ; lobular breast carcinoma in situ; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Ductal, Breast; Carcinoma, Lobular; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Partial Breast Re-Irradiation (Experimental): Partial Breast Re-Irradiation (PBrI) 3D-Conformal External Beam 1.5 Gy x 15 (BID) to 45 Gy Total
  Interventions: Radiation: 3D-Conformal External Beam

INTERVENTIONS:
Radiation: 3D-Conformal External Beam — Radiation was to be delivered in 2 fractions per day, each of 1.5 Gy, separated by at least six hours, given in 15 consecutive working days to a total of 30 fractions and 45 Gy. Radiation was to be prescribed to the treatment unit isocenter, positioned at the approximate center of the planning target volume.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Giving radiation therapy after surgery kill any remaining tumor cells and may be an effective treatment for breast cancer.

PURPOSE: This phase II trial is studying how well radiation therapy works in treating women with locally recurrent breast cancer previously treated with repeat breast-conserving surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate skin, breast, and chest wall adverse events occurring within 1 year after completion of 3D-conformal partial-breast re-irradiation following repeat breast-preserving surgery in patients with locally recurrent breast carcinoma.

Secondary

* To evaluate the adverse events occurring after 1 year from the completion of re-irradiation and at any time.
* To evaluate in-breast control rate in patients treated with this regimen.
* To evaluate freedom-from-mastectomy rate in these patients.
* To evaluate the rate of circulating tumor cells (CTCs) in this patient population and to document eradication of CTCs by locoregional therapy.
* To determine whether translational objective will correlate with eradication or presence of CTCs with in-breast recurrence and distant metastasis-free survival.
* To evaluate cosmesis as judged by the patient and independent evaluation.
* To evaluate distant metastasis-free survival, mastectomy-free survival, and overall survival of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients undergo 3-dimensional conformal accelerated partial-breast irradiation twice daily, 5 days a week, for 3 weeks.

Some patients undergo blood sample collection at baseline and within 3 weeks after completion of radiotherapy for circulating tumor cells analysis.

Some patients complete questionnaires on cosmesis at baseline and at 1 and 3 years following radiotherapy.

After completion of study therapy, patients are followed up periodically for 4-5 years and then every year thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally recurrent breast carcinoma consistent with the following cell types:

  * Invasive ductal breast carcinoma
  * Medullary ductal breast carcinoma
  * Tubular ductal breast carcinoma
  * Mucinous ductal breast carcinoma
  * Lobular breast carcinoma
  * Ductal carcinoma in situ (DCIS)

    * No Paget disease of the nipple
  * Target lumpectomy cavity must be clearly defined and the target lumpectomy cavity/ whole-breast reference volume must be < 30% based on a post-operative, pre-treatment CT scan
  * Tumor size ≤ 3 cm in greatest dimension on pathologic specimen
  * Negative histologic margins of resection and no tumor on ink following breast-preserving surgery of local recurrence (Re-excision is permitted to achieve negative margins)
  * Axilla negative or ≤ 3 positive lymph nodes without extracapsular extension
  * If the in-breast recurrence is DCIS and/or microinvasive disease, a sentinel lymph node (SLN) evaluation is not required, but if performed:
  * Patients with a negative sentinal lymph node (SLN) biopsy are eligible for enrollment
  * Patients with a positive SLN biopsy require an axillary lymph node (ALN) dissection (ALND is not required if the SLN is not identified)
  * Patient is eligible if 0-3 positive ALNs without extracapsular extension is documented
* If the in-breast recurrence is invasive disease and:

  * No prior ALN dissection or SLN dissection only:

    * Patient is required to undergo axillary evaluation with either a SLN or ALN dissection
    * If the SLN is not identified or if the SLN is positive for metastatic disease then an ALN dissection is required
    * Patient is eligible for enrollment if encounter 0-3 positive lymph nodes without extracapsular extension
  * • Prior ALN dissection: negative clinical exam: patient is eligible for enrollment

    * It is recommended, but not required, that the patient undergo ultrasound evaluation of the axilla and the lymph node draining regions of the breast; any suspicious areas are to be biopsied and if positive followed with an ALN dissection
    * Patient is eligible for enrollment if biopsies are negative or 0-3 axillary lymph nodes without extracapsular extension are encountered
  * Prior ALN dissection: positive clinical exam: biopsy required

    * If biopsy is negative, patient is eligible for enrollment
    * If biopsy is positive an ALN dissection is required
    * Patient is eligible for enrollment if biopsies are negative or 0-3 axillary lymph nodes without extracapsular extension encountered
* Ipsilateral breast mammogram and MRI within 120 days prior to study entry
* Contralateral breast mammogram within 12 months of study entry
* For invasive in-breast recurrence, no more than 120 days since whole-body (positron emission tomography) PET-CT scan OR CT scan of the chest, abdomen, and pelvis, and bone scan
* No multicentric ipsilateral breast recurrence or regional recurrence (other than axilla)
* Patients must have a breast technically amenable to partial-breast irradiation
* No metastatic disease documented by physical exam or radiographic evaluation (for patients with invasive disease)
* No skin involvement
* No prior contralateral mastectomy
* Estrogen and progesterone status must be known

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Menopausal status not specified
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other invasive malignancy within the past 3 years except ipsilateral breast cancer and/or nonmelanoma skin cancer
* No collagenous diseases, specifically systemic lupus erythematosus, scleroderma, or dermatomyositis
* No psychiatric or addictive disorders that would preclude obtaining informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 2 weeks since prior chemotherapy and recovered
* No concurrent intensity-modulated radiotherapy
* No concurrent chemotherapeutic agents, including trastuzumab

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-06; Primary Completion 2014-11 (Actual); Study Completion 2022-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas W. Arthur, MD, Principal Investigator — Massey Cancer Center
Locations (58):
- United States (57):
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Roy and Patricia Disney Family Cancer Center at Providence Saint Joseph Medical Center, Burbank, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - JFK Medical Center, Atlantis, Florida
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Tate Cancer Center at Baltimore Washington Medical Center, Glen Burnie, Maryland
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - St. Barnabas Medical Center Cancer Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - Highland Hospital of Rochester, Rochester, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan-Kettering Cancer Center - Rockville Centre, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Delaware County Regional Cancer Center at Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Cancer Care Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
- Cross Cancer Institute at University of Alberta, Edmonton, Alberta, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Partial Breast Re-Irradiation
Started | 65
Has Baseline PT QOL Data (Eligible patients who consented to QOL study & have patient-reported baseline data) | 46
Has Baseline MD QOL Data (Eligible patients who consented to QOL study & have physician-assessed baseline data) | 44
Has Baseline/12-month PT QOL Data (Eligible patients who consented to QOL study & have patient-reported baseline/12-month data) | 36
Has Baseline/12-Month MD QOL Data (Eligible patients who consented to QOL study & have physician-assessed baseline/12-month data) | 35
Has Baseline/36-month PT QOL Data (Eligible patients who consented to QOL study & have patient-reported baseline/36-month data) | 32
Has Baseline/36-Month MD QOL Data (Eligible patients who consented to QOL study & have physician-assessed baseline/36-month data) | 27
All Eligible Patients | 58
Completed | 58 (Subjects with data available for analysis are considered to have completed the study.)
Not Completed | 7
Not completed — Protocol Violation | 4
Not completed — No protocol treatment received | 3

BASELINE CHARACTERISTICS:
Population: All eligible patients
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
Age, Continuous [Median (Full Range); unit: years] | 67 [44 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3+ Treatment-related Skin, Fibrosis, and Breast Pain Adverse Events
Description: Adverse events (AEs) were graded with Common Terminology Criteria for Adverse Events (CTCAE) version 4. Grade refers to the severity of the AE. The Common Terminology Criteria for Adverse Events (CTCAE) v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. Based on a rate of 4% for the AEs of interest, a rate of ≥ 13% for these AEs with re-irradiation would be unacceptable. A sample size of 55 evaluable pts (eligible & started protocol treatment) would provide: 86% power to conclude an unacceptable rate of the specified AEs, if the true AE rate was at least 13%; 93% probability to not conclude an unacceptable rate of the specified AEs, if the true AE rate is 4%. If ≥ 5 pts have treatment-related AEs, then the treatment-related AE rate was considered unacceptable.
Time Frame: From the end of radiation to 1 year.
Population: The first 55 eligible patients who completed treatment and achieved 1 year of follow-up.
Measure: Number; unit: participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 55
participants | 1

2. Secondary Outcome: In-breast Recurrence
Description: The definition of treatment failure is histologic evidence of recurrent carcinoma, either invasive or non-invasive (except LCIS) in the ipsilateral breast. Clinical evidence of carcinoma by physical examination and/or mammograms and/or MRI will not be construed as evidence of treatment failure without biopsy proof but will be considered as suspicious for recurrence. Ipsilateral breast recurrences will be considered local (infield) if they occur within the prescription isodose volume; they will be considered peripheral if they occur between the prescription isodose volume and a volume 2 cm outside of the prescription isodose volume. Ipsilateral recurrences will be considered non-contiguous or extra field if they are beyond the peripheral volume described above.
Time Frame: From registration to date of recurrence or last follow-up. Analysis occurs after all patients have been potentially followed for 3 years.
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
percentage of participants | 3.7 [0.7 to 11.4]
Statistical Analysis 1: Comparison: Partial Breast Re-Irradiation; Assuming a 3-year rate of 25% using a chi-squared test, a sample size of 55 patients will ensure at least 90% probability of detecting a reduction in the 3-year ipsilateral in-breast recurrence rate from 25% to 9%, with a significance level of 0.05 (1-sided). In-breast recurrence will be estimated using the cumulative incidence method; Test type: Superiority or Other; p = 0.0002, Chi-squared

3. Secondary Outcome: Freedom From Mastectomy
Description: Failure is mastectomy of the treated breast. Mastectomy rate at 3 years is reported, using the cumulative incidence with death as competing risk. Mastectomy-free survival is reported in outcome measure 10.
Time Frame: From registration to date of mastectomy or last follow-up. Analysis occurs after all patients have been potentially followed for 3 years.
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
percentage of participants | 5.2 [1.3 to 13.1]

4. Secondary Outcome: Number of Patients With Detectable/Undetectable/Unevaluable Circulating Tumor Cells (CTCs)
Description: CTCs in peripheral blood were assessed using the CellSearch (trademark) system. A stringent algorithm was used to classify cell images as a CTC. A CTC must express EpCAM [epithelial cell adhesion molecule] and not leukocyte lineage-specific antigens, exhibit cytoplasmic expression of cytokeratin, and contain a nucleus that binds DAPI [4',6-doamidino-2-phenylindole]. A cell image is not a CTC if any of the previous criterion are missing. A subject is categorized as "Detectable" if the patient had a CTC and "Undetectable" if the subject had no CTCs. If neither category could be determined, then the subject was categorized as "Unevaluable."
Time Frame: Prior to the start of radiation and 3 weeks after last radiation treatment.
Population: Eligible patients who consented to participate in the CTC portion of the trial
Measure: Count of Participants; unit: Participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 47
Participants
  Pre-treatment: Detectable | 8
  Pre-treatment: Undetectable | 32
  Pre-treatment: Unevaluable | 7
  Post-treatment: Detectable | 8
  Post-treatment: Undetectable | 26
  Post-treatment: Unevaluable | 13

5. Secondary Outcome: Treatment-related Adverse Events (AEs) Any Time
Description: AEs were graded with Common Terminology Criteria for Adverse Events (CTCAE) version 4. Grade refers to the severity of the AE. The Common Terminology Criteria for Adverse Events (CTCAE) v4.0 assigns Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 1 Mild AE, Grade 2 Moderate AE, Grade 3 Severe AE, Grade 4 Life-threatening or disabling AE, Grade 5 Death related to AE. The overall highest grade for each patient was computed from all reported adverse events definitely, probably, or possibly related to protocol treatment.
Time Frame: From the end of radiation to end of follow-up. Will be evaluated at the time of the primary analysis.
Population: All eligible patients
Measure: Number; unit: percentage of participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
percentage of participants
  Grade 5 | 0
  Grade 4 | 0
  Grade 3 | 10.3
  Grade 2 | 32.8
  Grade 1 | 41.4

6. Secondary Outcome: Distant Metastasis-free Survival
Description: Failures are appearance of ipsilateral axillary, infraclavicular, internal mammary, or supraclavicular recurrences; distant metastases confirmed radiographically and/or pathologically; or death due to any cause. Note that a distant metastases was only considered a treatment failure if accompanied by an in-breast recurrence.
Time Frame: From registration to date of distant metastasis, death or last follow-up. Analysis occurs after all patient have been potentially followed for 3 years.
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
percentage of participants | 94.8 [84.8 to 98.3]

7. Secondary Outcome: Mastectomy-free Survival
Description: Failure is mastectomy of the treated breast or death due to any cause. Mastectomy-free survival rate at three years was estimated using the Kaplan-Meier method.
Time Frame: From registration to date of mastectomy, death or last follow-up. Analysis occurs after all patients have been potentially followed for 3 years.
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
percentage of participants | 89.7 [78.4 to 95.2]

8. Secondary Outcome: Overall Survival
Description: Failure is death due to any cause. Three-year overall survival rate was estimated using the Kaplan-Meier method.
Time Frame: From registration to date of death or last follow-up. Analysis occurs after all patients have been potentially followed for 3 years.
Population: All eligible patients.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
percentage of participants | 94.8 [84.8 to 98.3]

9. Secondary Outcome: Treatment-related Adverse Events Occurring After One Year From Completion of Re-irradiation
Description: AEs were graded with CTCAE version 4. The overall highest grade for each patient is computed from reported adverse events definitely, probably, or possibly related to protocol treatment occurring after one year from completion of re-irradiation.
Time Frame: After 1 year from the end of radiation.
Population: All eligible patients
Measure: Number; unit: percentage of participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 58
percentage of participants
  Grade 5 | 0
  Grade 4 | 0
  Grade 3 | 6.9
  Grade 2 | 22.4
  Grade 1 | 24.1

10. Secondary Outcome: Change in Patient-Reported Cosmetic Outcomes From Baseline to 12-Months as Measured by the Breast Cancer Treatment Outcome Scale (BCTOS)
Description: The Breast Cancer Treatment Outcome Scale (BCTOS) is a 22-item tool to assess cosmetic results using patient self-reports. This brief self-report instrument has high reliability and validity, and it has been used in a variety of previous studies on recovery from breast cancer treatment. It is comprised of three subscales (functional status, cosmetic status, and breast specific pain). Response options for each BCTOS item form a four-point Likert scale evaluating the differences between the treated and the untreated breast (1=no, 2=slight, 3=moderate, 4=large difference). The score for each subscale is the mean of the ratings over all items belonging to that specific subscale. Change was calculated as the value at 12 months minus the value at baseline. A positive change reflects a decline at 12 months and a negative change reflects an improvement at 12 months.
Time Frame: Baseline and 12 months from the start of radiation treatment.
Population: Eligible patients who consented to participate in the quality of life study and have baseline and 12-month BCTOS data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 36
units on a scale
  Functional status | 0.04 (0.41)
  Cosmetic | 0.09 (0.65)
  Breast-specific pain | -0.21 (0.62)
Statistical Analysis 1: Comparison: Partial Breast Re-Irradiation; Functional status; Test type: Other; Effect size = 0.10 — Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7
Statistical Analysis 2: Comparison: Partial Breast Re-Irradiation; Cosmetic; Test type: Other; Effect size = 0.14 — Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7
Statistical Analysis 3: Comparison: Partial Breast Re-Irradiation; Breast-specific pain; Test type: Other; Effect size = 0.34 — Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7

11. Secondary Outcome: Change in Patient-Reported Cosmetic Outcomes From Baseline to 36-Months as Measured by the Breast Cancer Treatment Outcome Scale (BCTOS)
Description: The Breast Cancer Treatment Outcome Scale (BCTOS) is a 22-item tool to assess cosmetic results using patient self-reports. This brief self-report instrument has high reliability and validity, and it has been used in a variety of previous studies on recovery from breast cancer treatment. It is comprised of three subscales (functional status, cosmetic status, and breast specific pain). Response options for each BCTOS item form a four-point Likert scale evaluating the differences between the treated and the untreated breast (1=no, 2=slight, 3=moderate, 4=large difference). The score for each subscale is the mean of the ratings over all items belonging to that specific subscale. Change was calculated as the value at 36 months minus the value at baseline. A positive change reflects a decline at 36 months and a negative change reflects an improvement at 36 months.
Time Frame: Baseline and 36 months from the start of radiation treatment.
Population: Eligible patients who consented to participate in the quality of life study and have baseline and 36-month BCTOS data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 32
units on a scale
  Functional status | -0.02 (0.47)
  Cosmetic | 0.19 (0.59)
  Breast-specific pain | -0.20 (0.72)
Statistical Analysis 1: Comparison: Partial Breast Re-Irradiation; Functional status; Test type: Other; Effect size = 0.04 — Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7
Statistical Analysis 2: Comparison: Partial Breast Re-Irradiation; Cosmetic; Test type: Other; Effect size = 0.32 — Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7
Statistical Analysis 3: Comparison: Partial Breast Re-Irradiation; Breast-specific pain; Test type: Other; Effect size = 0.28 — Effect sizes are interpreted as negligible: < 0.3; small: 0.3 to < 0.5; moderate: 0.5 to < 0.7; and large ≥ 0.7

12. Secondary Outcome: Number of Patients With Good/Excellent Cosmesis Using the NRG Oncology/Radiation Therapy Oncology Group (RTOG) Cosmetic Rating Scale
Description: Physicians rated cosmesis using a 4 point NRG Oncology/RTOG established criteria scale:
  Excellent - when compared to the untreated breast or the original appearance of the breast, there is minimal/no difference in the size or shape of the treated breast.
  Good - there is a slight difference in the size or shape of the treated breast as compared to the opposite breast or the original appearance of the treated breast.
  Fair - obvious differences in the size and shape of the treated breast. This change involves quarter or less of the breast.
  Poor - marked change in the appearance of the treated breast involving more than a quarter of the breast tissue.
Time Frame: Baseline,12, and 36 Months from the start of radiation treatment.
Population: Eligible patients who consented to participate in the quality of life study and have baseline data
Measure: Count of Participants; unit: Participants
Arm/Group | Partial Breast Re-Irradiation
Number analyzed (Participants) | 46
Participants
  Baseline-Excellent/Good: number analyzed (Participants) | 44
  Baseline-Excellent/Good | 26
  12-Month-Excellent/Good: number analyzed (Participants) | 35
  12-Month-Excellent/Good | 22
  36-Month-Excellent/Good: number analyzed (Participants) | 27
  36-Month-Excellent/Good | 14

13. Secondary Outcome: 12-Month BCTOS Mean Subscale Scores by 12-Month NRG Oncology/RTOG Cosmetic Rating Scale
Description: Patient-Reported BCTOS is comprised of 3 subscales (functional status, cosmetic status, breast specific pain). Responses for each item form a 4-point Likert scale evaluating the differences between the treated and untreated breast (1=no, 2=slight, 3=moderate, 4=large difference). Higher scores reflect poorer outcomes.
  Physicians rated cosmesis using a 4 point NRG Oncology/RTOG established criteria scale:
  Excellent - when compared to the untreated breast or the original appearance of the breast, there is minimal/no difference in the size or shape of the treated breast.
  Good - there is a slight difference in the size or shape of the treated breast as compared to the opposite breast or the original appearance of the treated breast.
  Fair - obvious differences in the size and shape of the treated breast. This change involves quarter or less of the breast.
  Poor - marked change in the appearance of the treated breast involving more than a quarter of the breast tissue.
Time Frame: 12 Months from the start of radiation treatment.
Population: Eligible patients who consented to participate in the quality of life study and have baseline and 12-month BCTOS data
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Functional Score: Patient-Reported: 12-Month Functional Score
- Cosmetic Score: Patient-Reported: 12-Month Cosmetic Score
- Breast-Specific Pain Score: Patient-Reported: 12-Month Breast-Specific Pain Score
Arm/Group | Functional Score | Cosmetic Score | Breast-Specific Pain Score
Number analyzed (Participants) | 32 | 32 | 32
units on a scale
  Physician 12-Month Score: Excellent: number analyzed (Participants) | 4 | 4 | 4
  Physician 12-Month Score: Excellent | 1.03 (0.06) | 1.67 (0.57) | 1.33 (0.47)
  Physician 12-Month Score: Good: number analyzed (Participants) | 15 | 15 | 15
  Physician 12-Month Score: Good | 1.14 (0.25) | 1.88 (0.44) | 1.53 (0.45)
  Physician 12-Month Score: Fair: number analyzed (Participants) | 11 | 11 | 11
  Physician 12-Month Score: Fair | 1.55 (0.53) | 2.19 (0.69) | 1.82 (0.77)
  Physician 12-Month Score: Poor: number analyzed (Participants) | 2 | 2 | 2
  Physician 12-Month Score: Poor | 1.06 (0.09) | 2.48 (1.21) | 2.50 (1.18)
Statistical Analysis 1: Comparison: Functional Score; Test type: Other; p = 0.054, Spearman rank-order correlation test
Statistical Analysis 2: Comparison: Cosmetic Score; Test type: Other; p = 0.044, Spearman rank-order correlation test
Statistical Analysis 3: Comparison: Breast-Specific Pain Score; Test type: Other; p = 0.087, Spearman rank-order correlation test

ADVERSE EVENTS:
Description: Subjects experiencing more than one of a given adverse event are counted only once for that adverse event.
Arm/Group | Partial Breast Re-Irradiation
Serious Adverse Events (participants affected / at risk) | 3/58
Other Adverse Events (participants affected / at risk) | 52/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Partial Breast Re-Irradiation (N=58)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
Multi-organ failure (General disorders) | 1
Pain (General disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin induration (Skin and subcutaneous tissue disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1
Lymphedema (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Partial Breast Re-Irradiation (N=58)
Anemia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 32
Localized edema (General disorders) | 8
Pain (General disorders) | 12
Skin infection (Infections and infestations) | 5
Dermatitis radiation (Injury, poisoning and procedural complications) | 17
Fracture (Injury, poisoning and procedural complications) | 3
Seroma (Injury, poisoning and procedural complications) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Fibrosis deep connective tissue (Musculoskeletal and connective tissue disorders) | 16
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 5
Superficial soft tissue fibrosis (Musculoskeletal and connective tissue disorders) | 19
Dizziness (Nervous system disorders) | 5
Insomnia (Psychiatric disorders) | 3
Breast atrophy (Reproductive system and breast disorders) | 13
Breast pain (Reproductive system and breast disorders) | 21
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 12
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 29
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Skin induration (Skin and subcutaneous tissue disorders) | 14
Telangiectasia (Skin and subcutaneous tissue disorders) | 11
Hot flashes (Vascular disorders) | 8
Hypertension (Vascular disorders) | 3
Lymphedema (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.